CLINICAL TRIAL: NCT03928899
Title: The Best Timing of Delivery in Women With GDM That is Controlled With Only Diet and Exercise
Brief Title: The Best Timing of Delivery in Women With GDM Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Wang Chen, Doctor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUFHIOL
Record Dates: First submitted 2019-04-18; First posted 2019-04-26 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Gestational Diabetes; Induction of Labor Affected Fetus / Newborn
Keywords: induction; caesarean section; fetal weight; Bishop score
MeSH Terms: conditions — Diabetes, Gestational; Fetal Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- old guideline group (No Intervention): Women randomized to the "old guideline group" will be followed up once-weekly by electronic fetal heart rate monitoring and biophysical profile until 40 weeks 0 days (unless a medical indication arises), when induction of labor was then offered.
- new procedure group (Experimental): Women randomized to "new procedure group" will first undergo fetal weight ultrasound estimation at 38 weeks 0 days to 38 weeks 6 days of gestation, if the fetus is estimated to be LGA/macrosomia by ultrasound, women should have an elective induction of labor immediately (at 38 weeks 0 days to 38 weeks 6 days of gestation). On the contrary, if the fetus is estimated to be normal size, the pregnant women were then given a cervical assessment. If the Bishop score ≥6, women will have at least weekly follow-up visits with their doctors and unless a medical indication is present, continue pregnancy and have selective induction at 40 weeks 0 days of gestation. Whereas, if the Bishop score <6, women will be followed up until 41 weeks 0 days of gestation with a close assessment of fetal wellbeing through the cardiotocographic trace. And women who will not deliver by this gestational age will be admitted for labor induction. Certainly, medical indication should warrant delivery without delay.
  Interventions: Procedure: New procedure

INTERVENTIONS:
Procedure: New procedure — An optimal management on the timing and mode of delivery of pregnant women with GDM, by a comprehensive assessment and consideration of their fetal weight, gestational age, and cervical ripeness.
  Other Names: New
  Arms: new procedure group

SUMMARY:
The investigatiors aimed to conduct a well-designed RCT to firstly focus on GDM women controlled with only diet and exercise, and provide an optimize process on their timing and mode of delivery

DETAILED DESCRIPTION:
GDM is a common complication of pregnancy and even mildly hyperglycemia could significantly affect fetal growth. Optimal delivery timing in women with GDM remains controversial. This decision process involves balancing the potential for complications that are caused by increased interventions with the benefit of avoidance of future adverse outcomes. Thus, the aim of the present trial is to explore the best management on the timing of delivery of pregnant women with GDM that controlled with only diet and exercise, which can both decrease the risk of macrosomia and the risk of cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women
* in vertex presentation
* GDM that is controlled with only diet and exercise
* at 37 weeks 0 days to 37 weeks 6 days of gestation
* more than 18 years old
* have no other contraindications to vaginal delivery.

Exclusion Criteria:

* prior caesarean section or myomectomy
* any known contraindications to vaginal delivery
* uncertain gestational age
* non reassuring foetal wellbeing necessitating delivery
* maternal pregnancy-related disease necessitating delivery (any hypertensive disorder, cardiac disease, renal insufficiency、immune diseases, et al.)
* placenta previa, accreta, vasa previa
* known foetal anomaly
* negative reproductive history
* ruptured membranes or known oligohydramnios (defined as AFI < 5 or MVP < 2 ) before 37weeks 6 days of gestation
* fetal growth restriction, defined as EFW < 10th percentile
* known HIV positivity because of modified delivery plan
* signs of labor (regular painful contractions with cervical change) before 37weeks 6 days of gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
caesarean section rate | 41weeks

SECONDARY OUTCOMES:
mode of delivery | 41weeks
  spontaneous or operative vaginal delivery, caesarean section；the investigator will use questionnaire to collect these information from their medical record
onset of labour | 41weeks
  spontaneous or instrumental third stage of labour, planned or emergency caesarean section;the investigator will use questionnaire to collect these information
operative vaginal delivery indication | 41weeks
  chorioamnionitis defined as a clinical diagnosis before delivery; fetal distress; arrest of second stage of labour; maternal complicatio;the investigator will use questionnaire to collect these information from their medical record
caesarean section indication | 41weeks
  induction failed; chorioamnionitis defined as a clinical diagnosis before delivery; fetal distress; arrest of second stage of labour; failed instrumental delivery; maternal complication; elective
method of induction of labour | 41weeks
  prostaglandin tablet regime; artificial rupture of amniotic membranes; oxytocin exclusive if used to accelerate normal labour
indication for induction | 41weeks
  randomised to treatment; prelabour rupture of membranes > 2 hours and no regular contractions; fetal growth restriction; reduced fetal movements/suspected fetal distress; pregnancy induced hypertension; pre-eclampsia/eclampsia; obstetric cholestasis;the investigator will use questionnaire to collect these information from their medical record
gestational age | 41weeks
intrapartum complications | 41weeks
  placental abruption; cord prolapse; postpartum haemorrhage defined as bleeding of 500/1000ml or more in the first 24 hours following the vaginal/ caesarean section delivery of the baby; third or fourth degree perineal laceration; admission to intensive care unit; hysterectomy; maternal venous thromboembolism
birth weight | 41weeks
neonatal sex | 41weeks
neonatal plasma glucose level collected 1-2h after delivery | 41weeks
neonatal hypoglycemia | 41weeks
stillbirth | 41weeks
  a baby delivered with no signs of life after24 completed weeks of pregnancy
shoulder dystocia | 41weeks
  the investigator will use questionnaire to collect these information from their medical record
death before discharge from hospital | 41weeks
Apgar at 1 min, Apgar at 5 min, Apgar at 10 minutes | 41weeks
cord blood artery pH | 41weeks
neonatal respiratory distress | 41weeks
  the investigator will use questionnaire to collect these information from their medical record
birth trauma | 41weeks
  subdural haematoma, intracerebral or intraventricular haemorrhage, spinal-cord injury, basal skull fracture, peripheral-nerve injury, long bone fracture
NICU admission | 41weeks
seizures | 41weeks
  the investigator will use questionnaire to collect these information from their medical record
hypotonia | 41weeks
  the investigator will use questionnaire to collect these information from their medical record
intubation and ventilation for > 24 h | 41weeks
oxygen required | 41weeks
the utilization of medical resources | 41weeks
  That includes: number of clinic visits post randomization to admission for delivery, number of times for having non-stress tests, ultrasounds and contraction stress tests, Use of induction and ripening agents, maximum dose of oxytocin, interval from randomization to delivery, number of hours on the labor and delivery unit, maternal postpartum length of hospital stay, neonatal length of hospital stay
the mothers' expectations and experience of childbirth | 41weeks
  measured by the Labour Agentry Scale (which is designed to assess the expectations and experiences of personal control during childbirth, with higher scores indicating greater perceived control during childbirth)
rate of labor pain | 41weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided